CLINICAL TRIAL: NCT05987202
Title: Impact of Postnatal Betamethasone Treatment on Closure of Ductus Arteriosus in Preterm Infants
Brief Title: Betamethasone and Closure of Ductus Arteriosus
Acronym: CELESTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0779
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Persistent Ductus Arteriosus
Keywords: Prematurity; Ductus arteriosus; Steroids; Betamethasone; Bronchopulmonary dysplasia
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants born between January 1st, 2018 and December 31st, 2022: All infants born alive before 37 weeks between January 1st, 2018 and December 31st, 2022 with PDA
  Interventions: Other: DA closure in a population of premature infants

INTERVENTIONS:
Other: DA closure in a population of premature infants — Evaluate the incidence of DA closure in a population of premature infants treated with BTM per os for bronchopulmonary dysplasia

SUMMARY:
The ductus arteriosus (DA) normally closes after birth as a result of exposure to oxygen. Its persistence of DA (PDA) occurs in 20 to 50% of very preterm infants and is associated with significant morbidity and mortality: prolongation of respiratory assistance, pulmonary haemorrhage, -necrotizing enterocolitis (NECU), intraventricular haemorrhage and death.

PDA management is one of the most discussed aspects in neonatology. The treatment is either conservative (controlled fluid intake, monitoring of cerebral flows, diuretics), or pharmacological (ibuprofen or paracetamol per os), or surgical (thoracotomy + ligature or catheterization + plug). The success rate of pharmacological treatment of CAP is 30% in the most immature children. When medical treatment fails, surgical or endovascular treatment is considered. However, these are associated with complications such as recurrent nerve lesion, thoracotomy, failure to close DA, migration of the plug. Therefore individualized assessment balances the expected benefits of CAP treatment against the risks associated with the treatments for each patient.

The main complication of CAP is the impossibility of weaning the patient from ventilatory assistance. On the one hand because of PDA, but also very often because of the concomitant development of bronchopulmonary dysplasia (BPD) due to pulmonary lesions secondary to assisted ventilation and especially to inflammation. At 3 weeks of life, if attempts at ventilatory weaning have failed, postnatal corticosteroid therapy is considered in the 4th week of life in accordance with current recommendations.

The most commonly used postnatal corticosteroids are dexamethasone (DXM), hydrocortisone hemisuccinate (HSHC) and betamethasone (BTM). DXM (intravenous) is effective and is the most widely used product worldwide, but its use is associated with impaired postnatal growth and suboptimal neurodevelopment. HSHC (intravenous) is an alternative to DXM and has shown some effectiveness, without the adverse effects of DXM. The BTM is also an alternative, but has been used less than the other products because it is not widely available in some countries. Its advantage is that it can be given orally, but there is little published data on the effect of BTM. In this context, it has been used in some neonatal units and have shown some effectiveness.

In the Neonatology department of the Croix Rousse hospital, oral BTM has been used since 2005 and has been evaluated favorably, since it allows the child to be weaned from ventilatory assistance. When using BTM, we observed not only a positive respiratory effect, but also DA closure, reducing the need for ligation of the ductus arteriosus by surgery or catheterization

ELIGIBILITY:
* Inclusion Criteria :

  * born between January 2018 and December 2022
  * at a gestational age below 37 weeks,
  * hospitalized in the Neonatal unit of Croix-Rousse hospital,
  * presenting a hemodynamically significant DA
  * treated by BTM for bronchopulmonary dysplasia
* Exclusion Criteria :

  * Children having closed their ductus arteriosus before administration of the betamethasone course
  * Children who died before or during treatment.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants born between january 2018 and December 2022, at a gestational age below 37 weeks, hospitalized in the Neonatal unit of Croix-Rousse hospital, presenting an hemodynamically significant DA and treated by BTM for bronchopulmonary dysplasia
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of children with favorable evolution of the CAP | through study completion, an average of 6 months
  Number of children with favorable evolution of the CAP Percentage of children who present a favorable evolution of the CAP defined as a closure of the CAP or a CAP which becomes hemodynamically insignificant, under the effect of treatment with BTM

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation néonatale - Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Derived] Remy A, Vincent M, Pastor-Diez B, Picaud JC. Late postnatal steroid treatment using oral betamethasone can help to close ductus arteriosus in extremely preterm infants who cannot be weaned from ventilation. Eur J Pediatr. 2024 Nov 28;184(1):50. doi: 10.1007/s00431-024-05840-9. PMID 39604779